CLINICAL TRIAL: NCT04718194
Title: Developing Efficient Intervention Technologies to Reduce Stigma-Related Stress, Mental Health Problems, and HIV Risk Among Young Chinese MSM
Brief Title: Developing Online Interventions to Reduce Stigma-Related Stress, Sexual Health, and HIV Risk Among Young Chinese MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Central South University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2000029433; 1R21TW011762-01 (NIH); 5R21TW011762-02 (NIH)
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: LGBTQ; Sexual Behavior; HIV Risk
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESTEEM iCBT (Experimental): The online CBT treatment consists of 10 weekly modules that participants will complete over the course of 10 weeks.
  Interventions: Behavioral: ESTEEM iCBT
- Self-monitoring (Placebo Comparator): Participants will be asked to indicate their past 7-day mood; stress experiences; and mental and behavioral health on an online survey experience once per week for 10 weeks
  Interventions: Behavioral: Self-monitoring control

INTERVENTIONS:
Behavioral: ESTEEM iCBT — The online CBT treatment consists of 10 weekly modules that participants will complete over the course of 10 weeks.
  Arms: ESTEEM iCBT
Behavioral: Self-monitoring control — Participants will be asked to indicate their past 7-day mood; stress experiences; and mental and behavioral health on an online survey experience once per week for 10 weeks
  Arms: Self-monitoring

SUMMARY:
This study is a 2-arm RCT that will assess the efficacy of a culturally adapted, 10-session SGM-affirmative, internet-based cognitive behavioral therapy (iCBT) among young men who have sex with men (YMSM) in Hunan province China. The affirmative treatment called ESTEEM is based on a minority stress-focused, CBT framework. In collaboration with colleagues at Central South University (CSU), the investigators will assess whether a culturally adapted version of iCBT ESTEEM demonstrates significant reductions in HIV risk behavior and mental health symptoms (e.g., depression, anxiety) compared to self-monitoring of stress and mood.

DETAILED DESCRIPTION:
The primary objective is to evaluate the preliminary efficacy of a Chinese-adapted version of iCBT ESTEEM on YMSM's sexual health and HIV risk behavior. The secondary objectives of this study are to determine whether iCBT ESTEEM impacts HIV/sexually transmitted infections (STI) results and symptoms of depression and anxiety, as well as whether baseline minority stress exposure moderates treatment efficacy, such that participants with the most minority stress exposure benefit more from iCBT ESTEEM than those in the self-monitoring of stress and mood condition.

The proposed prospective study will follow a 2-arm RCT design where 120 Chinese YMSM participants will be randomly assigned to one of two conditions:

1. ESTEEM iCBT: This online CBT treatment consists of 10 weekly modules that participants will complete over the course of 10 weeks. Modules contain weekly psychoeducational text and vignettes about minority stress and mental health; brief videos illustrating the CBT skills; and homework exercises that therapists review and provide feedback on. Homework exercises include weekly tracking of stress and mood, practicing new skills (e.g., mindfulness, cognitive restructuring), and exercises related to considering the origins of stress and negative emotions that participants may be experiencing. Therapists provide feedback after each homework assignment, including reviewing each participant's treatment goals as part of the first session's homework. Therapists who support this condition will be instructed to incorporate SGM-specific content and feedback into homework reviews. In the US, modules were adapted directly from the in-person materials (e.g., therapist manual, participant handouts) used in our previously successful trials of this treatment. The treatment has also been recently culturally adapted for in-person treatment among Chinese YMSM and found to be acceptable and feasible.
2. Self-monitoring control: In this control condition, participants will be asked to indicate their past 7-day mood, stress experiences, and mental and behavioral health on an online survey. This type of self-monitoring has been shown to yield improvement in behavioral health outcomes. Self-reporting SGM stress experiences has also been shown to produce reductions in depression symptoms over time. Participants will record these experiences once per week for 10 weeks.

Before the full trial is launched, the investigators will ensure comprehension of the ESTEEM iCBT online module material with 10 separate YMSM, as well as gather their feedback on the usability of the iCBT online platform.

ELIGIBILITY:
Inclusion Criteria:

* 16-30 years old
* Live in Hunan province China
* Current gender identity as male
* Report past 12-month sex with men
* Be confirmed HIV-negative upon at-home testing
* Report past 3-month condomless/PrEP-less anal sex
* Past-week symptoms of depression or anxiety using the Brief Symptom Inventory-4 cutoff of 2.5 on either the depression subscale, anxiety subscale, or both
* No past 3-month mental health services of more than 2 visits per month
* Weekly access to internet on a laptop, desktop, or tablet device
* Ability to read, write, and speak in Mandarin
* Provision of informed consent

Exclusion Criteria:

* Current active suicidality or homicidality (defined as active intent or concrete plan, as opposed to passive ideation)
* Evidence of active and untreated mania or psychosis that could interfere with the participant's ability to volitionally consent to research or interfere with their ability to safely and reliably complete research

Ages: 16 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, Ph.D., Principal Investigator — Yale University
Locations (1):
- Central South University, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 12 months after study completion for three years.
Access Criteria: Data access requests from qualified academic investigators for non-commercial research interests will be reviewed by study investigators. Requestors will be required to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via online and paper advertisements on social networking platforms and in the lobbies of LGBTQ+ friendly organizations. 425 prospective participants completed the initial online screener.
Pre-assignment Details: All 120 participants who completed consent and were enrolled logged into the iCBT platform, completed the baseline survey, and were randomized.
Period: Overall Study
Arm/Group | ESTEEM iCBT | Self-monitoring
Started | 60 | 60
Completed ≥ 1 Module of the Intervention | 58 | 60
Completed 4-month Follow-up | 54 | 60
Completed 8-month Follow-up | 54 | 60
Completed | 54 | 60
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESTEEM iCBT | Self-monitoring | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.73 (3.36) | 22.72 (3.09) | 23.22 (3.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 60 | 60 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Han nationality | 58 | 55 | 113
  Ethnicity: Hmong/Miao minority | 2 | 1 | 3
  Ethnicity: Tujia minority | 0 | 3 | 3
  Ethnicity: Hui minority | 0 | 1 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Gay/homosexual | 57 | 53 | 110
  Bisexual | 3 | 7 | 10
Education Degree [Count of Participants; unit: Participants]
  Junior high school or less | 0 | 1 | 1
  High school/vocational school | 9 | 6 | 15
  College/four-year university | 44 | 47 | 91
  Graduate school or above | 7 | 6 | 13
Marital/Relationship Status [Count of Participants; unit: Participants]
  Single, without a regular partner | 22 | 24 | 46
  Single, but having regular partner | 34 | 33 | 67
  Married | 2 | 3 | 5
  Divorced | 2 | 0 | 2
Estimated Income Per Month [Count of Participants; unit: Participants]
  <3000RMB | 30 | 29 | 59
  3000-5000 | 14 | 17 | 31
  5000-800 | 9 | 8 | 17
  >8000RMB | 7 | 6 | 13
Employment Status [Count of Participants; unit: Participants]
  Full-time job | 26 | 29 | 55
  Part-time job | 5 | 4 | 9
  Student | 26 | 24 | 50
  Unemployed | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Past 90-Day Condomless Anal Sex Acts
Description: The Timeline Follow-Back (TLFB) assesses retrospective estimates of HIV-related sexual behavior in the past 30 days. The TLFB was originally developed in interview format, but has been adapted as online self-report questionnaire. Participants report on daily partner type (e.g. main, casual), type of sexual behavior (e.g. insertive anal sex, receptive anal sex, oral sex), and condom use. The TLFB has good test-retest reliability, convergent validity, and agreement with collateral reports for HIV-related sexual behavior. Administration time ranges from 10-30 minutes.
  For this primary outcome measure, condomless anal sex (CAS) with main or casual partners will be determined. The primary comparison will be change in the number of CAS acts from baseline to 8 months post-baseline.
Time Frame: Baseline, 4 months, 8 months
Population: Intent to Treat Population (participants analyzed according to their original treatment assignment regardless of adherence to protocol) for all participants who completed 4/8-month follow-up assessments.
Measure: Mean (Standard Deviation); unit: condomless anal sex acts
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
condomless anal sex acts
  Baseline | 1.98 (3.78) | 1.80 (2.34)
  4-Month Post-Baseline | 0.58 (1.06) | 0.80 (2.04)
  8-Month Post-Baseline | 0.50 (1.22) | 0.65 (1.36)

2. Secondary Outcome: Change in Number of Past 90-Day Condomless Anal Sex Acts With Casual Partners
Description: The Timeline Follow-Back (TLFB) assesses retrospective estimates of HIV-related sexual behavior in the past 30 days. The TLFB was originally developed in interview format, but has been adapted as online self-report questionnaire. Participants report on daily partner type (e.g. main, casual), type of sexual behavior (e.g. insertive anal sex, receptive anal sex, oral sex), and condom use. The TLFB has good test-retest reliability, convergent validity, and agreement with collateral reports for HIV-related sexual behavior. Administration time ranges from 10-30 minutes.
  For this secondary outcome measure, condomless anal sex (CAS) with casual partners only will be determined.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: condomless anal sex acts
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
condomless anal sex acts
  Baseline | .58 (0.98) | 0.50 (1.40)
  4-Month Post-Baseline | .11 (0.42) | 0.22 (0.67)
  8-Month Post-Baseline | 0 (0.00) | 0.08 (0.46)

3. Secondary Outcome: Change in Depression
Description: Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). A sum score of 9 items indicates depression severity, with higher scores indicating higher severity and a scores ranging from 0-27. A 10th item indicates functional impairment. A cutoff score of 7 or more indicates high likelihood of a depressive episode.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
units on a scale
  Baseline | 12.40 (5.70) | 10.40 (5.28)
  4-Month Post-Baseline | 8.33 (3.85) | 10.00 (4.74)
  8-Month Post-Baseline | 7.28 (4.47) | 10.00 (3.98)

4. Secondary Outcome: Change in Anxiety
Description: Anxiety will be measured using the Generalized Anxiety Disorder-7 scale (GAD-7). A sum score of 7 items indicates anxiety severity, with higher scores indicating higher severity and scores ranging from 0 to 21. An 8th item indicates functional impairment. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate, and severe anxiety, respectively.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
units on a scale
  Baseline | 9.55 (5.05) | 9.03 (5.06)
  4-Month Post Baseline | 5.72 (3.77) | 8.80 (4.64)
  8-Month Post Baseline | 5.54 (3.34) | 8.47 (4.22)

5. Secondary Outcome: Change in Disordered Alcohol Use
Description: Disordered alcohol use will be assessed using the Alcohol Use Disorders Identification (AUDIT) instrument. The AUDIT consists of 10 items. Items 1 to 9 are scored 0, 1, 2, 3, or 4, and item 10 is scored 0, 2, or 4. Higher scores indicate greater alcohol use, with scores ranging from 0 to 40. Total scores of 8 or more are recommended as indicators of hazardous and harmful alcohol use, as well as possible alcohol dependence.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
units on a scale
  Baseline | 4.32 (5.47) | 4.88 (5.87)
  4-Month Post-Baseline | 3.44 (4.57) | 4.68 (5.53)
  8-Month Post-Baseline | 2.43 (3.52) | 5.30 (5.89)

6. Secondary Outcome: Change in Disordered Drug Use
Description: Disordered drug use other than alcohol will be assessed using the Drug Use Disorders Identification (DUDIT) instrument. The DUDIT consists of 11 items. Items 1 to 9 are scored 0, 1, 2, 3, or 4, and items 10 and 11 are scored 0, 2, or 4. Higher scores indicate greater drug use, with scores ranging from 0 to 44. A score of 25 points or more is recommended as an indicator of drug dependence.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
units on a scale
  Baseline | 1.38 (2.99) | 1.97 (3.82)
  4-Month Post-Baseline | 0.91 (2.17) | 1.40 (3.03)
  8-Month Post-Baseline | 0.61 (1.39) | 1.33 (2.91)

7. Secondary Outcome: Change in Suicidal Ideation
Description: Suicidal ideation will be measured using the Suicidal Ideation Attributes Scale (SIDAS). Total SIDAS scores are calculated as the sum of the five items, with controllability (item 2) reverse scored (10=0, 9=1, …, 0=10). Higher scores indicate greater suicidality, with total scores ranging from 0 to 50.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
units on a scale
  Baseline | 5.07 (6.70) | 5.47 (7.36)
  4-Month Post-Baseline | 2.09 (4.56) | 4.17 (7.30)
  8-Month Post-Baseline | 1.76 (3.74) | 2.97 (6.10)

8. Secondary Outcome: Change in Concealment Motivation
Description: Motivation to conceal sexual minority identity will be assessed using the Concealment Motivation subscale of the Lesbian, Gay, and Bisexual Identity Scale (LGBIS). The three subscale items, rated on a 6-point scale, will be averaged for a total score, ranging from 1 to 6. Higher scores indicate higher concealment motivation.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 4.66 (1.27) | 4.36 (1.25)
  4-Month Post-Baseline | 4.59 (1.23) | 4.40 (1.25)
  8-Month Post-Baseline | 4.55 (1.23) | 4.44 (1.22)

9. Secondary Outcome: Change in Acceptance Concerns
Description: Acceptance concerns of sexual minority identity will be assessed using the Acceptance Concerns subscale of the Lesbian, Gay, and Bisexual Identity Scale (LGBIS). The three subscale items, rated on a 6-point scale, will be averaged for a total scores ranging from 1 to 6. Higher scores indicate higher acceptance concerns.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 4.73 (1.23) | 4.63 (1.05)
  4-Month Post-Baseline | 4.38 (1.18) | 4.75 (1.05)
  8-Month Post-Baseline | 4.36 (1.40) | 4.53 (1.11)

10. Secondary Outcome: Change in Internalized Homonegativity
Description: Internalized homonegativity will be assessed using the Internalized Homophobia subscale of the Lesbian, Gay, and Bisexual Identity Scale (LGBIS). The three subscale items, rated on a 6-point scale, will be averaged for a total scores, ranging from 1 to 6. Higher scores indicate higher internalized homonegativity.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 3.68 (1.60) | 3.19 (1.30)
  4-Month Post-Baseline | 3.60 (1.52) | 3.37 (1.46)
  8-Month Post-Baseline | 3.30 (1.59) | 3.22 (1.37)

11. Secondary Outcome: Change in Emotion Dysregulation
Description: Emotion dysregulation will be assessed using the 18-item Difficulties in Emotion Regulation Scale-Short Form (DERS-SF). Items are rated on a 5-point scale from 1-5; items 1, 4, and 6 are reverse coded. Items are summed for a total score, ranging from 18 to 90, where higher scores indicate higher emotion dysregulation.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 55.9 (9.64) | 54.7 (10.7)
  4-Month Post-Baseline | 50.0 (11.5) | 55.2 (10.0)
  8-Month Post-Baseline | 48.2 (10.6) | 53.0 (10.2)

12. Secondary Outcome: Change in Perceived Social Support
Description: Perceived social support will be measured using the 12-item Multidimensional Scale of Perceived Social Support (MPSS). Items are rated on a 7-point scale from 1-7 and averaged for a total score, ranging from 1 to 7, with higher scores indicating higher perceived social support.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 3.53 (1.28) | 3.66 (1.30)
  4-Month Post-Baseline | 3.79 (1.34) | 3.49 (1.26)
  8-Month Post-Baseline | 3.98 (1.30) | 3.81 (1.18)

13. Secondary Outcome: Change in Rumination
Description: Rumination will be measured using the 5-item Brooding Subscale of the Ruminative Responses Scale (RRS). Items are rated on a 4-point scale from 1-4 and summed for a total scores, ranging from 5 to 20, with higher scores indicating higher rumination.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 13.9 (3.33) | 14.2 (3.13)
  4-Month Post-Baseline | 12.6 (3.12) | 13.6 (3.67)
  8-Month Post-Baseline | 12.3 (2.77) | 13.0 (3.48)

14. Secondary Outcome: Change in HIV/STI Testing
Description: The Past 4-month HIV/STI Testing Questionnaire consists of 7 multiple choice questions previously developed by the study PI for another study asking participants about their HIV/STI testing history. The questionnaire consists of questions, such as, "Have you provided a urine sample as part of any STI test in the last 4 months" with response options of "yes," "no," or "I don't remember." Scores were coded with "yes" being 1 and "no" being 0, and and a total score was assessed as the average of all scores. Thus, total scores ranged from 0 to 1, with higher scores indicating greater HIV/STI testing in the past 4 months.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 0.850 (.360) | 0.867 (.343)
  4-Months Post-Baseline | 0.815 (.392) | 0.883 (.321)
  8-Months Post-Baseline | 0.870 (.339) | 0.900 (0.303)

15. Secondary Outcome: Change in Condom Use
Description: The Decisional Balance for Condom Use Scale is an 18-item psychometrically validated scale measuring one's motivation to increase condom use (e.g., "I would feel bad if my friends found out I had sex without a condom"), with response options ranging between 1 = not at all to 5 = extremely. Scores are summed for a total scores, ranging from 18 to 90, with lower scores are indicative of greater likelihood to use a condom.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 61.2 (8.29) | 61.5 (10.4)
  4-Month Post-Baseline | 59.1 (9.65) | 60.6 (9.99)
  8-Month Post-Baseline | 57.4 (8.04) | 59.3 (10.0)

16. Secondary Outcome: Change in Safer Sex
Description: The Safer Sex Questionnaire is a psychometrically validated measure and consists of 13-items based on a 5-point Likert scale assessing one's confidence in avoiding having anal sex without a condom in various contexts. Scores are summed for a total score, ranging from 13 to 65, with higher scores are indicative of greater safer sex self-efficacy.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 55.5 (9.46) | 55.9 (9.63)
  4-Months Post-Baseline | 56.5 (8.50) | 57.1 (9.95)
  8-Months Post-Baseline | 58.8 (7.05) | 57.9 (8.53)

17. Secondary Outcome: Change in HIV Test Results
Description: Participants will be provided with self-administered rapid HIV testing kits at baseline and 8-months post-baseline to assess for incidence of HIV.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
Participants
  Baseline: Positive | 0 | 0
  Baseline: Negative | 54 | 60
  4-Month Post-Baseline: Positive | 0 | 0
  4-Month Post-Baseline: Negative | 54 | 60
  8-Month Post-Baseline: Positive | 0 | 0
  8-Month Post-Baseline: Negative | 54 | 60

18. Secondary Outcome: Change in Syphilis Test Results
Description: Participants will be provided with self-administered rapid syphilis testing kits at baseline and 8-months post-baseline to assess for incidence of syphilis.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
Participants
  Baseline: Positive | 0 | 1
  Baseline: Negative | 54 | 59
  4-Month Post-Baseline: Positive | 0 | 1
  4-Month Post-Baseline: Negative | 54 | 59
  8-Month Post-Baseline: Positive | 0 | 1
  8-Month Post-Baseline: Negative | 54 | 59

19. Other Pre Specified Outcome: Change in Depression Severity
Description: As an exploratory outcome, depression severity will be measured using the Overall Depression Severity & Impairment Scale (ODSIS). This 5 item measure uses a 0-4 rating scale and sums across the items for a total score ranging from 0 to 20. Higher scores indicate greater severity of depression.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 7.80 (4.15) | 7.03 (3.45)
  4-Months Post-Baseline | 4.70 (3.15) | 6.45 (4.02)
  8-Months Post-Baseline | 3.80 (2.68) | 5.32 (3.24)

20. Other Pre Specified Outcome: Change in Anxiety Severity
Description: As an exploratory outcome, anxiety severity will be measured by the Overall Anxiety Severity & Impairment Scale (OASIS). This 5 item measure uses a 0-4 rating scale and sums across the items for a total score ranging from 0 to 20. Higher scores indicate greater severity of anxiety.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 9.10 (3.23) | 8.80 (3.06)
  4-Months Post-Baseline | 5.78 (2.66) | 7.57 (3.59)
  8-Months Post-Baseline | 5.19 (2.39) | 6.82 (2.63)

21. Other Pre Specified Outcome: Change in Self-Esteem
Description: As an exploratory outcome, self-esteem will be measured using the 10-item Rosenberg Self-Esteem Scale. Items are rated on a 4 point scale from 0-3; items 4, 6, 9, 10, and 11 are reverse scored. Items are summed for a total score ranging from 0 to 30, where a higher score indicates greater self-esteem.
Time Frame: Baseline, 4 months, 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM iCBT | Self-monitoring
Number analyzed (Participants) | 54 | 60
score on a scale
  Baseline | 25.3 (5.46) | 25.9 (4.90)
  4-Months Post-Baseline | 27.2 (4.60) | 25.7 (4.45)
  8-Months Post-Baseline | 27.9 (4.66) | 25.4 (4.48)

ADVERSE EVENTS:
Time Frame: Up to 8 months
Arm/Group | ESTEEM iCBT | Self-monitoring
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
This trial was conducted during the COVID-19 pandemic and associated restrictive policies in China, which might have influenced intervention efficacy in ways unknown, although stress, mental health, and behavioral outcomes such as HIV-transmission-risk behavior have all been documented to have been influenced by the pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT04718194/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04718194/SAP_001.pdf
  • Informed Consent Form (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT04718194/ICF_003.pdf